CLINICAL TRIAL: NCT00100295
Title: Controlled Trial of an Herbal Treatment for Juvenile Attention Deficit Hyperactivity Disorder
Brief Title: Herbal Treatment for Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K23AT000929 (NIH)
Record Dates: First submitted 2004-12-28; First posted 2004-12-29 (Estimated); Last update posted 2007-10-26 (Estimated); Status verified 2007-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Adolescent; Child; Phytotherapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Hypericum extract LI 160

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Herbal treatment
  Interventions: Drug: Hypericum perforatum
- B (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hypericum perforatum — 300 mg capsule taken three times a day
  Other Names: St. John's Wort
  Arms: A
Other: Placebo — 300 mg given three times a day, containing rice protein powder
  Arms: B

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of an herbal product for the treatment of attention deficit hyperactivity disorder (ADHD) in children and adolescents.

DETAILED DESCRIPTION:
ADHD is a common childhood disorder associated with concentration problems and disruptive behavior. Evidence suggests that herbal remedies may be as effective as standard drug therapies in treating ADHD symptoms. This study will determine the safety and efficacy of an herbal treatment in children and adolescents with ADHD.

This study will last 9 weeks. Participants will be randomly assigned to receive either an herbal product or placebo three times a day for the duration of the study. Participants will come in for weekly study visits at which their ADHD symptoms and any side effects will be assessed by self-report rating scales.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD
* Score of greater than 1.5 standard deviation above the age and gender norms on the ADHD-IV rating scale
* Parents and children can understand English
* Parents and children willing to attend all study visits
* Able to swallow study medication
* Willing to use acceptable methods of contraception

Exclusion Criteria:

* Severe depression
* History of bipolar disorder, psychosis, severe conduct disorder, or other serious medical conditions
* Use of medications that may interact with the herbal product
* Current use of medications to treat ADHD
* Previous use of Hypericum
* Pregnancy

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2005-02; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
ADHD-IV rating scale | Difference between baseline and end of study
side effects scale | Freqency of events during entire study

SECONDARY OUTCOMES:
Child Behavior Checklist, Youth Self Report Form | Baseline and end of study

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Weber, ND, MPH, Principal Investigator — Bastyr University
Locations (1):
- Bastyr University, Kenmore, Washington, United States

REFERENCES:
- [Derived] Weber W, Vander Stoep A, McCarty RL, Weiss NS, Biederman J, McClellan J. Hypericum perforatum (St John's wort) for attention-deficit/hyperactivity disorder in children and adolescents: a randomized controlled trial. JAMA. 2008 Jun 11;299(22):2633-41. doi: 10.1001/jama.299.22.2633. PMID 18544723